CLINICAL TRIAL: NCT01128387
Title: A Phase I/II Study of Panitumumab/Cisplatin/Fluorouracil Combined With Radiation Preoperatively for Patients With Locally Advanced Esophageal Cancer
Brief Title: Trial of Panitumumab/Cisplatin/Fluorouracil Combined With Radiation in Esophageal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2009-0214; RO09211 (Other: University of Wisconsin Carbone Cancer Center); NCI-2011-00735 (Registry Identifier: NCI Trial ID); A533300 (Other: UW Madison); SMPH\HUMAN ONCOLOGY\HUMAN ONCO (Other: UW Madison)
Record Dates: First submitted 2010-05-17; First posted 2010-05-21 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2018-03

CONDITIONS: Cancer
Keywords: esophageal cancer; Locally advanced esophageal cancer
MeSH Terms: conditions — Neoplasms; Esophageal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dose Level -1 (Experimental): Panitumumab/Cisplatin/Fluorouracil and Radiation therapy 1.5mg/kg Panitumumab, 60mg/m2 cisplatin, 750mg/m2 5FU (Fluorouracil)
  Interventions: Drug: Panitumumab
- Dose Level 1 (Experimental): Panitumumab/Cisplatin/Fluorouracil and Radiation therapy 1.5mg/kg Panitumumab, 80mg/m2 cisplatin, 1000mg/m2 5FU (Fluorouracil)
  Interventions: Drug: Panitumumab

INTERVENTIONS:
Drug: Panitumumab — dose escalating 1.5mg/kg or 2.5mg/kg weekly during radiation. Cisplatin on Days 1 and 29, Fluorouracil on Days1-4 and Days 29-32.

SUMMARY:
The overall study objective is to evaluate the dose limiting toxicities and the recommended phase II dose of Panitumumab when combined with the standard of care treatment with cisplatin, fluorouracil and radiation in patients with locally advanced esophageal cancer. The investigators will also be assessing the ability of PET (Positron Emission Tomography) imaging to predict the degree of pathologic response.

All patients will have a pre-study FDG (F-18 Fluorodeoxyglucose) PET scan and will receive radiation therapy and chemotherapy over a 35 day period. 4-8 weeks post radiation and chemotherapy patients will be restaged with a PET/CT scan. It is anticipated that approximately 30 patients enrolled will undergo an esophagectomy which is considered standard of care post radiation and chemotherapy. The surgery will allow us to compare this study regimen to the historical standard of care (Cisplatin/fluorouracil chemotherapy with radiation therapy).

ELIGIBILITY:
Inclusion Criteria:

1. Locally Advanced Esophageal cancer (stages T1N1 or T2-4 any N)
2. Histology must be adenocarcinoma or squamous cell carcinoma
3. Must be surgical candidate based on evaluation by a thoracic surgeon
4. must have adequate organ function as defined by routine lab tests

Exclusion Criteria:

1. Insitu carcinoma
2. prior chemotherapy for esophageal cancer
3. Metastatic (stage IV disease)
4. Tumors <5cm from the cricopharyngeus muscle, Tumors with >75% of tumor located within the stomach
5. Active, uncontrolled cardiac disease
6. subjects with >Grade 2 neuropathies. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Ritter, M.D., Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the University of Wisconsin Hospital and Clinics between 2010 and 2013.
Groups:
- Dose Level 1: Panitumumab/Cisplatin/Fluorouracil and Radiation therapy Panitumumab: dose escalating 1.5mg/kg or 2.5mg/kg weekly during radiation. Cisplatin on Days 1 and 29, Fluorouracil on Days1-4 and Days 29-32.
  1.5mg/kg Panitumumab,80mg/m2 cisplatin, 1000mg/m2 5FU (Fluorouracil)
- Dose Level -1: Panitumumab/Cisplatin/Fluorouracil and Radiation therapy Panitumumab: dose escalating 1.5mg/kg or 2.5mg/kg weekly during radiation. Cisplatin on Days 1 and 29, Fluorouracil on Days1-4 and Days 29-32.
  1.5mg/kg Panitumumab,60mg/m2 cisplatin, 750mg/m2 5FU
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level -1
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1: Panitumumab/Cisplatin/Fluorouracil and Radiation therapy Panitumumab: dose escalating 1.5mg/kg or 2.5mg/kg weekly during radiation. Cisplatin on Days 1 and 29, Fluorouracil on Days1-4 and Days 29-32.
  1.5mg/kg Panitumumab,80mg/m2 cisplatin, 1000mg/m2 5FU
- Dose Level -1: Panitumumab/Cisplatin/Fluorouracil and Radiation therapy Panitumumab: dose escalating 1.5mg/kg or 2.5mg/kg weekly during radiation. Cisplatin on Days 1 and 29, Fluorouracil on Days1-4 and Days 29-32.
  1.5mg/kg Panitumumab, 60mg/m2 cisplatin, 750mg/m2 5FU
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level -1 | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 3 | 5
Age, Continuous [Mean (Full Range); unit: years] | 60.3 [51 to 69] | 62.6 [53 to 69] | 61.5 [51 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: MTD of Panitumumab in Combination With Cisplatin/Fluorouracil and Radiation for Locally Advanced Esophageal Cancer Determined by Number of Participants Experiencing DLT
Description: Maximum Tolerated Dose (MTD) will be where 0 of 6 patients experienced Dose Limiting Toxicities (DLT) from start until 28 days after the completion of radiation. The investigator considered DLTs related to the treatment to be: grade 4 hematologic toxicity, grade 3 hematologic toxicity lasting >7 days, any neutropenic fever, all grade 3 non-hematologic toxicities (excluding alopecia and nausea/vomiting/diarrhea if controlled with antiemetics or anti-diarrheal agents), grade 4 lab abnormality (whether symptomatic or asymptomatic), any treatment related to death, any toxicity associated with 1) any single interruption of radiation >10 treatment days, 2) >2 interruptions of radiation per course, 3) a delay in completion of radiation by >14 days beyond planned treatment schedule, 4) inability to deliver >80% of planned treatment doses, 5) any infield grade 4 toxicity
Time Frame: approximately 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level -1
Number analyzed (Participants) | 5 | 6
Participants | 2 | 0
Statistical Analysis 1: Comparison: Dose Level 1 vs Dose Level -1; Dose of Pantiumumab (in combination with Cisplatin & Fluorouracil - see below); Test type: Other; Maximum Tolerated Dose = 1.5
Statistical Analysis 2: Comparison: Dose Level 1 vs Dose Level -1; Dose of Cisplatin; Test type: Other; Maximum Tolerated Dose = 60
Statistical Analysis 3: Comparison: Dose Level 1 vs Dose Level -1; Dose of Fluorourcil; Test type: Other; Maximum Tolerated Dose = 750

2. Secondary Outcome: Pathologic Response
Description: From therapy initiation through 30 days post surgery. 5.5 weeks of XRT/chemo, 4-8weeks post Radiation (XRT)/Chemo subjects to undergo a surgical resection, and study will be completed 4 weeks post surgery with surgical morbidity and mortality information
Time Frame: 20 weeks.
Population: Data was not collected or analyzed for the pathologic response outcome measure.
Arm/Group | Dose Level 1 | Dose Level -1
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for up to 6 years, 3 months.
Description: Adverse events were collected at weekly visits.
Arm/Group | Dose Level 1 | Dose Level -1
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/5 | 2/6
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=5) | Dose Level -1 (N=6)
Alanine Amiotransferase (ALT) (General disorders) | 1 | 0
Aspartate Aminotransferase (AST) (General disorders) | 1 | 0
Bilirubin (General disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Conduction (Cardiac disorders) | 1 | 0
Dehydration (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hemorrhage (Gastrointestinal disorders) | 2 | 0
Infection (Infections and infestations) | 1 | 0
Leukocytes (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Platelets (Blood and lymphatic system disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Supraventricular and nodal arrhythmia (Cardiac disorders) | 0 | 1
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=5) | Dose Level -1 (N=6)
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Platelets (Blood and lymphatic system disorders) | 2 | 4
Leukocytes (Blood and lymphatic system disorders) | 3 | 6
Neutrophils (ANC (Absolute Neutrophil Count)) (Blood and lymphatic system disorders) | 3 | 1
Hemoglobin (Blood and lymphatic system disorders) | 5 | 3
Lymphopenia (Blood and lymphatic system disorders) | 4 | 2
Fatigue (General disorders) | 3 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Rash - Maculopapular (Skin and subcutaneous tissue disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 5
Mucositis (Gastrointestinal disorders) | 2 | 4
Esophagitis (Gastrointestinal disorders) | 5 | 0
Dehydration (Gastrointestinal disorders) | 1 | 5
Diarrhea (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Thrush (Gastrointestinal disorders) | 0 | 2
Dysgeusia (Gastrointestinal disorders) | 0 | 2
Belching (Gastrointestinal disorders) | 0 | 1
Mouth sores (Gastrointestinal disorders) | 0 | 1
Weight loss (Gastrointestinal disorders) | 0 | 2
Anorexia (Gastrointestinal disorders) | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 0 | 1
Creatinine (Metabolism and nutrition disorders) | 2 | 2
Hypoamagnesemia (Metabolism and nutrition disorders) | 2 | 2
Low sodium (hyponatremia) (Metabolism and nutrition disorders) | 3 | 2
Low calcium (hypocalcemia) (Metabolism and nutrition disorders) | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2
Neuropothy (Nervous system disorders) | 1 | 0
Depression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Pain (General disorders) | 2 | 0
Nocturia (Renal and urinary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The Standard of Care changed during this protocol, and the protocol was terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes